CLINICAL TRIAL: NCT00588718
Title: A Biologic Sample Study for the Validation of Biomarkers of Progressive NEC & Sepsis
Brief Title: A Biologic Validation of Biomarkers of Progressive NEC & Sepsis
Acronym: NEC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: R. Lawrence Moss (Other)
Collaborators: Mallinckrodt (Industry); Stanford University (Other); Baylor College of Medicine (Other); Johns Hopkins University (Other); University of Pennsylvania (Other); Yale University (Other)
Responsible Party: Sponsor-Investigator, R. Lawrence Moss, Surgeon In Chief, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: 26128
Record Dates: First submitted 2008-01-03; First posted 2008-01-09 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Necrotizing Enterocolitis
Keywords: Necrotizing enterocolitis; Progressive necrotizing enterocolitis; Proteomics in blood; Genomics in blood; Multi-center
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Infants who meet the entry criteria
- Controls: Banked blood samples from newborns who do not meet inclusion criteria for this study will be held at Stanford University Core Laboratory and will constitute controls. Proteomic and genomic profiles in blood samples of cases will be compared with blood samples of controls.

SUMMARY:
Necrotizing enterocolitis (NEC) is a severe, sometimes life-threatening inflammation of the intestine that occurs most often in premature babies. If it progresses, the wall of the intestine may perforate, spilling bacteria and stool into the abdomen. Parts or all of the intestine may die. Despite 30 years of clinical studies, the cause of NEC remains unknown.

In this study, we will be conducting an independent case-control validation study to verify the diagnostic and prognostic biomarker panels, develop validated biomarkers on boisensors in preparation for prospective validation studies, and conduct independent prospective validation of biosensor based biomarker panels on clinical samples.

ELIGIBILITY:
Inclusion Criteria - NEC/Sepsis Cohort GA < 29 weeks Current age equal or <12 weeks Suspicion of NEC or Sepsis

Exclusion - NEC/Sepsis Cohort Current or prior diagnosis of NEC Early onset infection (equal or <72 hours of life) Previous diagnosis of sepsis within 7 days Previous abdominal surgery Significant congenital anomaly

Inclusion Criteria - SIP Cohort Infants born at <29 weeks gestation Equal to or <12 weeks of age at the time of eligibility assessment a decision to perform surgery (or drain) for suspected NEC or SIP

Exclusion - SIP Cohort Congenital infection (Equal to <72 hours of life) Prior episode of NEC or SIP Prior laparotomy or drain for SIP or NEC

Ages: 72 Hours to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prematurely-born infants with with suspected necrotizing enterocolitis, sepsis or SIP who meet study entry criteria
Sampling Method: Non-Probability Sample
Enrollment: 740 (Estimated)
Dates: Start 2007-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To verify the diagnostic and prognostic biomarker panels with sufficiently powered new cohorts. | 4 years
  Study has been amended/extended. Test the NEC diagnostic panel for its ability to distinguish NEC from SIP. Develop validated biomarkers on biosensors in preparation for prospective validation studies.
  Independent prospective validation of biosensor based biomarker panels.

CONTACTS AND LOCATIONS:
Overall Officials: R. Lawrence Moss, MD, Principal Investigator — Nationwide Children's Hospital, The Ohio State University
Locations (1):
- R. Lawrence Moss, MD, Nationwide Children's Hospital, The Ohio State University, Karl Sylvester, MD, Stanford University, Stanford, Califorinia, Columbus, Ohio, United States

REFERENCES:
- [Result] Moss RL, Kalish LA, Duggan C, Johnston P, Brandt ML, Dunn JC, Ehrenkranz RA, Jaksic T, Nobuhara K, Simpson BJ, McCarthy MC, Sylvester KG. Clinical parameters do not adequately predict outcome in necrotizing enterocolitis: a multi-institutional study. J Perinatol. 2008 Oct;28(10):665-74. doi: 10.1038/jp.2008.119. Epub 2008 Sep 11. PMID 18784730